CLINICAL TRIAL: NCT00264615
Title: An Open-label, Double Conversion Study to Characterize the Pharmacokinetics of Lamotrigine When Switching Patients With Epilepsy on LAMICTAL Immediate-release to Extended-release Formulation and Vice Versa
Brief Title: Patients With Epilepsy Taking LAMICTAL Immediate-Release Who Switch To Extended-Release Formulation And Vice Versa
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Purpose: Treatment
Other Study IDs: LEP103944
Record Dates: First submitted 2005-12-09; First posted 2005-12-13 (Estimated); Last update posted 2016-09-23 (Estimated); Status verified 2016-09

CONDITIONS: Epilepsy
Keywords: once daily dosing; seizure; pharmacokinetics; epilepsy
MeSH Terms: conditions — Epilepsy; Seizures

INTERVENTIONS:
Drug: lamotrigine extended-release

SUMMARY:
Pharmacokinetic (PK) study to characterize changes in serum concentrations in epilepsy patients when switching from LAMICTAL immediate-release to extended-release and vice versa.

ELIGIBILITY:
Inclusion criteria:

* Confident diagnosis of epilepsy.
* Currently on LAMICTAL and up to 2 concomitant AEDs (anti-epileptic drugs).

Exclusion Criteria:

* Females of childbearing potential cannot be on hormonal contraceptives or hormone replacement therapy.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 45
Dates: Start 2005-10; Primary Completion 2006-06 (Actual); Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
Steady state AUC(0-24), Cmax and Ct (approximate Cmin) of lamotrigine

SECONDARY OUTCOMES:
Tmax and fluctuation index of lamotrigine
Adverse events, changes in blood pressure and heart rate
Change in seizure frequency during each of the study phases
Subject preference at End of Baseline and Extended-Release Treatment Phases

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (11):
- United States (11):
  - GSK Investigational Site, Anniston, Alabama
  - GSK Investigational Site, Sun City, Arizona
  - GSK Investigational Site, Lexington, Kentucky
  - GSK Investigational Site, Boston, Massachusetts
  - GSK Investigational Site, Reno, Nevada
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Toledo, Ohio
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Nashville, Tennessee
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Tompson DJ, Ali I, Oliver-Willwong R, Job S, Zhu L, Lemme F, Hammer AE, Vuong A, Messenheimer JA. Steady-state pharmacokinetics of lamotrigine when converting from a twice-daily immediate-release to a once-daily extended-release formulation in subjects with epilepsy (The COMPASS Study). Epilepsia. 2008 Mar;49(3):410-7. doi: 10.1111/j.1528-1167.2007.01274.x. Epub 2007 Sep 6. PMID 17825077
- [Derived] van Dijkman SC, de Jager NCB, Rauwe WM, Danhof M, Della Pasqua O. Effect of Age-Related Factors on the Pharmacokinetics of Lamotrigine and Potential Implications for Maintenance Dose Optimisation in Future Clinical Trials. Clin Pharmacokinet. 2018 Aug;57(8):1039-1053. doi: 10.1007/s40262-017-0614-5. PMID 29363050
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Annotated Case Report Form: LEP103944 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: LEP103944 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: LEP103944 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: LEP103944 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: LEP103944 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: LEP103944 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: LEP103944 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register